CLINICAL TRIAL: NCT01014377
Title: Assessment of the Safety of the VascuActive™ Device and Its Preliminary Efficacy on Foot Perfusion, Hemodynamics and Exercise Capacity in Patients With Peripheral Vascular Disease and Limb Ischemia
Brief Title: Effect of VascuActive Device on Foot Perfusion, Hemodynamics and Exercise Capacity in Patients With PVD & Limb Ischemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VascuActive LTD (Industry)
Responsible Party: Yuval Avni, VascuActive LTD
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VAS-01
Record Dates: First submitted 2009-11-11; First posted 2009-11-17 (Estimated); Last update posted 2010-05-21 (Estimated); Status verified 2010-05

CONDITIONS: Peripheral Vascular Diseases
MeSH Terms: conditions — Peripheral Vascular Diseases

INTERVENTIONS:
Device: VascuActive

SUMMARY:
The purpose of this study is to assess the safety and the immediate effect of the VascuActive device on patients with peripheral vascular disease and limb ischemia.

ELIGIBILITY:
Inclusion Criteria:

* Leg Ischemia, Fontaine grade IIa and IIb, i.e.: pain free walking distance in the range of 50 - 100 meters.
* Absent pulses in the two foot arteries (Anterior Tibial a., Posterior Tibial a.)
* ABI < 0.7 by Doppler, in at least one of the two foot arteries

Exclusion Criteria:

* Absent femoral pulses
* Venous insufficiency by Duplex
* Pregnancy
* Infectious disease
* Malignant disease
* Severe cardiac disease, e.g., CHF grade 3 or higher
* Acute MI within last 3 months
* CABG within last 3 months
* Other severe systemic disease

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Pain-free and Maximal walking distance | 1 hour

SECONDARY OUTCOMES:
Skin temperature | 1 hour
Skin blood flow | 1 hour
Transcutaneous partial pressure of O2 and CO2 | 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Asaf Harofe Medical Center, Zrifin, Israel